CLINICAL TRIAL: NCT05380752
Title: EXPANDED ACCESS PROTOCOL FOR TREATMENT OF INDIVIDUALS FOLLOWING EXPOSURE TO ORTHOPOX VIRUSES WITH TPOXX IV (TECOVIRIMAT INJECTION, 10 mg/mL)
Brief Title: Tecovirimat Intravenous Treatment for Orthopox Virus Exposure
Acronym: TPOXX IV
Status: No longer available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: SIGA Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: S-21-04; M-10922 (Other: USAMRDC)
Record Dates: First submitted 2022-04-27; First posted 2022-05-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Orthopox Virus Infection
MeSH Terms: interventions — tecovirimat

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: TPOXX IV (Tecovirimat Injection, 10 mg/mL) — IV solution (10 mg/mL) must be diluted with 2 parts 0.9% normal saline or 5% dextrose solution prior to dosing. Once diluted, the drug product should be stored at 2-8°C (36-46°F) and used as soon as possible (i.e., not more than 24 hours after dilution). Given via an IV infusion pump over a 6 hour period, twice daily, and for up to 7 days, or until the physician determines oral TPOXX may be given

SUMMARY:
* To provide a therapeutic option for patients not able to take the oral formulation of TPOXX (e.g., cannot swallow, vomiting) and who have confirmed or suspected (based on clinical signs and symptoms with known exposure while laboratory confirmation may be pending) orthopox virus infections OR who have a significant vaccinia adverse reaction (as defined in the protocol) resulting from vaccinia vaccination, secondary transmission, or other exposure;
* To collect data on the safety of TPOXX IV (tecovirimat injection, 10 mg/mL).

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed or suspected (based on clinical signs and symptoms with known or suspected exposure and/or positive or pending laboratory confirmation) orthopox virus infection.

   Note: Patients with a negative orthopox virus diagnostic test but with epidemiological and clinical evidence of an orthopox viral infection, especially those with evidence of clinical disease progression, may be included. Primary/Treating physician may consult with sponsor's Subject Matter Expert; OR Have developed a significant vaccinia adverse reaction (e.g., eczema vaccinatum, progressive vaccinia, generalized vaccinia that is severe or persistent, and select cases of inadvertent inoculation due to severe pain related to mucosal involvement, ocular involvement) resulting from vaccination, secondary transmission, or other exposure;
2. Be DoD-affiliated personnel (including active and reserve component service members, US civilian employees, contractors, other US personnel, and dependents, as well as allied military forces and local nationals) who have been granted access to the medical facility;
3. Unable to take the oral formulation of TPOXX (e.g., unable to swallow capsules or take medication powder dissolved in soft food or liquid, vomiting);
4. Is available for clinical follow-up for duration of the treatment and follow-up period;
5. Females of childbearing potential must use a highly effective method of contraception during treatment and for 30 days after the last dose of drug. Male patients with a female partner of childbearing potential must use an acceptable method of contraception and refrain from donating sperm during treatment and for 30 days after the last dose.

Exclusion Criteria:

1. Hypersensitivity to tecovirimat;
2. Unable or unwilling to cooperate with the requirements of the protocol;
3. Breastfeeding women: Nursing mothers will be counseled that tecovirimat has not been studied in breast-feeding women. Women who choose to continue breastfeeding will not be enrolled in this protocol. However, if a patient elects to stop breastfeeding for the duration of the study until 30 days after the last dose of the TPOXX IV, she may be enrolled.

Sex: All
Age Groups: Child, Adult, Older Adult